CLINICAL TRIAL: NCT05910073
Title: Efficacy Assessment of Lamina Curved Plate in Managing Oroantral Communication (OACs)
Acronym: CBSL
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0623
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-07

CONDITIONS: Oroantral Fistula
Keywords: Oroantral Fistula; Lamina Curved plate; Oral Surgery; Chronic sinusitis
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lamina curved plate: Use of a Lamina Curved plate (Osteobiol® Laboratory) in the treatment of OAC
  Interventions: Device: Lamina curved plate

INTERVENTIONS:
Device: Lamina curved plate — Use of a Lamina Curved plate (Osteobiol® Laboratory) in the treatment of OAC

SUMMARY:
The aim of this study is to assess the success rate, of using a Lamina Curved plate (Osteobiol® Laboratory) in the treatment of persistent OACs over 5mm.

DETAILED DESCRIPTION:
Oroantral communication (OAC) is an abnormal opening that forms between the maxillary sinus and oral cavity. This communication can occur as a result of tooth extraction, maxillofacial surgery or dental infections. Microorganisms from the oral cavity can then colonise the maxillary sinuses, leading to infections. Prompt and effective management of a OAC is essential to prevent complications such as acute or chronic sinusitis, facial pain or inflammation. Closure is usually made surgically with a local flap such as Fat pad flap, palatal or vestibular flap or with natural or synthetic biomaterials.

However, OACs may persist even after attempted closure, and there is also a risk of facial nerve damage during the dissection of the Bichat's flap.

All these factors prompt the evaluation of surgical procedures employed in the treatment of OACs, including the use of the Lamina Curved biomaterial from Osteobiol®. This biomaterial comprises a decalcified flexible plate made of heterologous cortical bone. It serves to reconstruct the sinus floor and isolate the sinus from the oral cavity. The plate is secured using osteosynthesis screws and possesses the characteristic of being resorbable.

The objective of this study is to investigate the success rate, of utilizing the Lamina Curved plate (Osteobiol® Laboratory) and to provide surgeons with an additional reference technique for treating OACs larger than 5mm.

ELIGIBILITY:
Inclusion Criteria :

* All patients with persistent OAC greater than 5mm treated with the use of an Osteobiol® Lamina curved plate
* Age ≥ 18 years
* Patients informed of the study and who did not object.

Exclusion Criteria :

* Follow-up less than 1 month after surgery
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major patients with persistent SBC greater than 5mm treated with an Osteobiol® Lamina curved plate.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment of Lamina Curved Plate in Managing Oroantral Communication | At the end of the study, an average of one month
  Number of patients with clinical closure of the OAC at D30 after the operation.

SECONDARY OUTCOMES:
Assessment of the complication rate | At the end of the study, an average of one month
  The complication rate of the technique will be evaluated by the number of patients having had at least one complication from D7 post-op to D30 post-op out of the number of patients included
Assessment of the rate of suture disunion | At the end of the study, an average of one month
  The rate of suture disunion will be assessed by the number of patients with at least one suture disunion from postoperative day 7 to postoperative day 30 out of the number of patients included

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nicolas Jaballah Magdeleine, Principal Investigator — Hôpital NOVO
Locations (1):
- Department of Stomatology - Hôpital NOVO Pontoise site, Pontoise, France

REFERENCES:
- [Background] Shahrour R, Shah P, Withana T, Jung J, Syed AZ. Oroantral communication, its causes, complications, treatments and radiographic features: A pictorial review. Imaging Sci Dent. 2021 Sep;51(3):307-311. doi: 10.5624/isd.20210035. Epub 2021 Jul 13. PMID 34621658
- [Background] Scott P, Fabbroni G, Mitchell DA. The buccal fat pad in the closure of oro-antral communications: an illustrated guide. Dent Update. 2004 Jul-Aug;31(6):363-4, 366. doi: 10.12968/denu.2004.31.6.363. PMID 15376721
- [Background] Lee JJ, Kok SH, Chang HH, Yang PJ, Hahn LJ, Kuo YS. Repair of oroantral communications in the third molar region by random palatal flap. Int J Oral Maxillofac Surg. 2002 Dec;31(6):677-80. doi: 10.1054/ijom.2001.0209. PMID 12521329
- [Background] Di Carlo R, Zara S, Ventrella A, Siani G, Da Ros T, Iezzi G, Cataldi A, Fontana A. Covalent Decoration of Cortical Membranes with Graphene Oxide as a Substrate for Dental Pulp Stem Cells. Nanomaterials (Basel). 2019 Apr 12;9(4):604. doi: 10.3390/nano9040604. PMID 31013705
- [Background] Caballe-Serrano J, Munar-Frau A, Delgado L, Perez R, Hernandez-Alfaro F. Physicochemical characterization of barrier membranes for bone regeneration. J Mech Behav Biomed Mater. 2019 Sep;97:13-20. doi: 10.1016/j.jmbbm.2019.04.053. Epub 2019 May 4. PMID 31085456
- [Background] Rossi R, Rancitelli D, Poli PP, Rasia Dal Polo M, Nannmark U, Maiorana C. The use of a collagenated porcine cortical lamina in the reconstruction of alveolar ridge defects. A clinical and histological study. Minerva Stomatol. 2016 Oct;65(5):257-68. PMID 27580650